CLINICAL TRIAL: NCT00001771
Title: I-123 Beta-CIT SPECT Studies of Dopamine and Serotonin Transporters in Neuropsychiatric Patients and Normal Volunteers
Brief Title: I-123 Brain Studies of Serotonin Metabolism in Psychiatric Patients and Normal Volunteers
Status: Completed | Type: Observational
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 980094; 98-M-0094
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2003-05

CONDITIONS: Healthy; Mental Disorder; Obsessive Compulsive Disorder; Schizophrenia; Tourette Syndrome
Keywords: Receptors; Re-Uptake; Neurotransmitters; Neuroimaging; Drug Abuse; Serotonin; Brain Scan; Tourette's Syndrome; Obsessive Compulsive Disorder; Schizophrenia; Normal Volunteer
MeSH Terms: conditions — Mental Disorders; Obsessive-Compulsive Disorder; Schizophrenia; Tourette Syndrome; Substance-Related Disorders

SUMMARY:
Abnormalities in the re-uptake of dopamine and serotonin have been described in various neuropsychiatric disorders and substance abuse. [I-123] Beta-CIT is a recently developed radioligand for SPECT imaging of dopamine and serotonin transporters. [I-123]Beta-CIT SPECT has been used at the SPECT-lab of the Clinical Brain Disorders Branch in over fifty subjects without adverse events. Due to the trace concentrations used, a pharmacological effect of Beta-CIT is unlikely and has not been observed. The purpose of this study is to use Beta-CIT and SPECT to study the expression of dopamine and serotonin transporters in vivo in normal controls and various patient populations to address hypothesized abnormalities of the transporters in different disorders and to understand the effects of genetic variations in the genes of these transporters on their in vivo expression.

DETAILED DESCRIPTION:
Abnormalities in the re-uptake of dopamine and serotonin have been described in various neuropsychiatric disorders and substance abuse. [I-123] Beta-CIT is a recently developed radioligand for SPECT imaging of dopamine and serotonin transporters. [I-123]Beta-CIT SPECT has been used at the SPECT-Lab of the Clinical Brain Disorders Branch in over fifty subjects without adverse events. Due to the trace concentrations used, a pharmacological effect of Beta-CIT is unlikely and has not been observed. The purpose of this study is to use Beta-CIT and SPECT to study the expression of dopamine and serotonin transporters in vivo in normal controls and various patient populations to address hypothesized abnormalities of the transporters in different disorders and to understand the effects of genetic variations in the genes of these transporters on their in vivo expression.

ELIGIBILITY:
INCLUSION CRITERIA:

No Axis I or Axis II diagnoses.

EXCLUSION CRITERIA FOR ALL SUBJECTS:

If the pregnancy test is positive or if the woman has reason to believe she might be pregnant, she will be excluded from this study.

Women who are breastfeeding will be excluded from this study to avoid unwarranted risk to their children.

Subjects with a prior reaction to iodine, iodine compounds, or shellfish will be excluded from this study.

Subjects with a history of thyroid disease or dysfunction will be excluded from this study.

Subjects with a history of recent substance abuse will be excluded from this study.

Subjects with metal objects in their bodies as specified in our MRI protocol (91-M-0124) will be excluded from this study.

If a structural abnormality of the brain is detected on MRI, subjects will be excluded from the study.

EXCLUSION CRITERIA FOR NORMAL CONTROLS:

Subjects with an Axis I or Axis II disorder will be excluded.

Subjects with concomitant medical or neurological disorders which require ongoing medication, or which may affect the central nervous system will be excluded.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 112
Dates: Start 1998-05; Study Completion 2003-05

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Mental Health (NIMH), Bethesda, Maryland, United States

REFERENCES:
- [Background] Bogerts B, Hantsch J, Herzer M. A morphometric study of the dopamine-containing cell groups in the mesencephalon of normals, Parkinson patients, and schizophrenics. Biol Psychiatry. 1983 Sep;18(9):951-69. PMID 6640008
- [Background] Czudek C, Reynolds GP. [3H] GBR 12935 binding to the dopamine uptake site in post-mortem brain tissue in schizophrenia. J Neural Transm. 1989;77(2-3):227-30. doi: 10.1007/BF01248935. PMID 2760605
- [Background] Innis RB, Seibyl JP, Scanley BE, Laruelle M, Abi-Dargham A, Wallace E, Baldwin RM, Zea-Ponce Y, Zoghbi S, Wang S, et al. Single photon emission computed tomographic imaging demonstrates loss of striatal dopamine transporters in Parkinson disease. Proc Natl Acad Sci U S A. 1993 Dec 15;90(24):11965-9. doi: 10.1073/pnas.90.24.11965. PMID 8265656